CLINICAL TRIAL: NCT02179632
Title: Disclosure of Industry Payments to Physicians and the Patient-Doctor Relationship
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Alison Hwong, MD-PhD Student, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB13-0727
Record Dates: First submitted 2014-06-26; First posted 2014-07-02 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Patient Doctor Trust
Keywords: disclosure; conflicts of interest; trust; patient doctor relationship

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Disclosure intervention zero (Experimental): Treatment Group 1: This group will be directed to ProPublica's Dollars For Docs physician payment disclosure registry for State of Massachusetts, and be asked to search for Dr. A. Participants will be asked to complete a worksheet reporting the total dollar amount listed for Dr. A, according to manufacturer, in 2012. Dr. A will be a physician the researchers have chosen who does not appear on the website and therefore did not receive any payments in 2012. Participants should report $0/not listed as the response. Following this stage, participants will be told that Dr. A does not appear on the website and therefore did not receive any payments.
  Interventions: Behavioral: Exposure to disclosure website
- Disclosure intervention low (Experimental): Treatment Group 2: This group will be directed to ProPublica's Dollars For Docs physician payment disclosure registry for State of Massachusetts, and be asked to search for Dr. B. Participants will be asked to complete a worksheet reporting the total dollar amount listed for Dr. B, according to manufacturer, in 2012. Dr. B will be a physician the researchers have chosen who received an aggregate amount that is a "low payment" (below $100) in 2012. Participants should report the dollar amount listed as the response. Following this stage, participants will be told the exact dollar amount for payments received by Dr. B in 2012.
  Interventions: Behavioral: Exposure to disclosure website
- Disclosure intervention high (Experimental): Treatment Group 3: This group will be directed to ProPublica's Dollars For Docs physician payment disclosure registry for State of Massachusetts, and be asked to search for Dr. C. Participants will be asked to complete a worksheet reporting the total dollar amount listed for Dr. C, according to manufacturer, in 2012. Dr. C will be a physician the researchers have chosen who received an aggregate amount that is a "high payment" (above $250) in 2012. Participants should report the dollar amount listed as the response. Following this stage, participants will be told the exact dollar amount for payments received by Dr. C in 2012.
  Interventions: Behavioral: Exposure to disclosure website
- Control group (No Intervention): Control Group: The control group will not be exposed to the disclosure website, but will participate in another online information-seeking task. These participants will visit the Farmer's Almanac website and be asked to search for temperature reports.

INTERVENTIONS:
Behavioral: Exposure to disclosure website — Participants are exposed to a physician payment disclosure website.
  Arms: Disclosure intervention high; Disclosure intervention low; Disclosure intervention zero

SUMMARY:
Pharmaceutical and medical device manufacturers work closely with doctors and hospitals, and the companies often pay large sums for consulting and advising services. Recipients of these payments and companies have stated that these financial relationships contribute to innovation in health care. However, multiple studies have also found that such payments have the potential to bias prescribing and treatment behaviors, and thus may lead to increases in health care costs.

One way to address potential conflicts of interest in medicine is public disclosure. As part of the Affordable Care Act, the Physician Payment Sunshine Act (PPSA) will establish a national disclosure website that posts all payments from pharmaceutical, medical device, and biologics manufacturers to doctors and hospitals starting in 2014. Payments exceeding $10 must be reported, and they will be listed by category, such as speaking engagements, meals, travel, and consulting services.

The Centers for Medicare and Medicaid Services (CMS) explicitly state in their Final Regulations for the PPSA that the disclosure website "will permit patients to make better informed decisions when choosing health care professionals and making treatment decisions," but the ways in which patients will evaluate and interpret disclosure remain unclear. One prominent topic in the discussion of disclosure is patient trust in health care providers and how transparency will affect the patient-doctor relationship-and, consequently, how the new law may affect physicians and hospitals.

DETAILED DESCRIPTION:
Patient trust is associated with improved self-care among patients with conditions from diabetes mellitus to HIV, and patient trust has also been found to correlate with medication adherence and continuity with physician. Therefore, an exploration of how large-scale public disclosure of payments will affect patient trust in doctors and the medical profession can help predict the effect of the policy on patient care.

Past studies of patient responses to disclosure present contradictory findings: some patients may refuse to see doctors who accept payments, while others may see the potential for conflicts of interest as only a small factor in the choice of physician. In one literature review, both patients and participants believed that disclosure would lead to increased confidence in their providers' decisions. Yet another study found that while disclosure does not have much impact on a person's willingness to participate in research, 59% of participants said that disclosure did not change their trust in the researcher or institution and 36% of participants indicated that their trust decreased. Moreover, in a role-playing experiment, patients who heard a disclosure statement said they would feel uncomfortable turning down a doctor's recommendations for fear of suggesting that the doctor was corrupt. However, none of these studies explicitly measured trust in a clinical relationship in the context of large-scale disclosure, which will be the setting for the PPSA website.

Defining Trust Both in the medical context and beyond, many definitions of trust have been proposed, and multiple measurement tools have been developed. Trust is generally thought of as "the willingness of a party to be vulnerable to the actions of another party based on the expectation that the other will perform a particular action important to the trustor, irrespective of the ability to monitor or control that other party." One of the most comprehensive conceptual models for trust in physicians and medical institutions is based on 5 dimensions: 1) fidelity, pursuing a patient's best interests; 2) competence, avoiding mistakes and producing the best results; 3) honesty, or telling the truth, 4) confidentiality, protection of private information, and 5) global trust, a holistic aspect.

There are multiple predictions for how disclosure will influence patient-provider relations when considering these dimensions. For example, the increased transparency about ties to industry could increase patient perceptions of honesty. Physicians who receive payments for consulting may be viewed as experts in their fields, and therefore may be seen as more competent. Alternatively, patients may question the fidelity of a doctor who receives payments, wondering if she has the patient's best interests as her priority. Thus, the implications for a national disclosure website on patient trust in physicians and the institution of medicine are unclear, despite CMS' claims that the PPSA will aid consumer decision-making. This project sets out to explore the effects of disclosure on patient trust in doctors and the medical profession.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be over 18 years of age, English-speaking, reside in Massachusetts, and have had an appointment with a physician within the last calendar year. These criteria will demonstrate a baseline level of interaction with the health care system. Our project uses data from health care professionals in Massachusetts, so we only wish to include people who live in Massachusetts.

Exclusion Criteria:

* Individuals under 18 years of age, non-English-speaking, who do not live in Massachusetts, and who have not had at least 1 appointment with a physician in the last calendar year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Trust-individual physician | Immediately after tasks are completed, 1-hour total
  This study will use the 10-item Wake Forest University Interpersonal Physician Trust Scale, rated on a 5-point Likert scale.
Trust-medical profession | Immediately after tasks are completed, 1-hour total
  This study will use the 10-item Patient Trust in the Medical Profession Scale, rated on a 5-point Likert scale.
Trust-industry | Immediately after tasks are completed, 1-hour total
  This study will an adapted 9-item Trust in Industry scale, rated on a 5-point Likert scale.

SECONDARY OUTCOMES:
Patient trust in own physician | Immediately after tasks are completed, 1-hour total
  Participants rate trust in own doctor on abbreviated 5-item interpersonal physician trust scale, rated on 5-point Likert scale.
Willingness to see doctor for care | Immediately after tasks are completed, 1-hour total
  Participants rate willingness to see physician for care, given disclosed payments, on 5-point Likert scale.
Change in trust score between rounds | Difference in scoring after 1st and 2nd round of tasks, 1 hour long total
  Difference between trust scores for 1st doctor vs. second doctor.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa S Lehmann, MD, PhD, Principal Investigator — Harvard Medical School, Partners Healthcare

REFERENCES:
- [Derived] Hwong AR, Sah S, Lehmann LS. The Effects of Public Disclosure of Industry Payments to Physicians on Patient Trust: A Randomized Experiment. J Gen Intern Med. 2017 Nov;32(11):1186-1192. doi: 10.1007/s11606-017-4122-y. Epub 2017 Jul 17. PMID 28717899